CLINICAL TRIAL: NCT02850692
Title: Portal Hypertension and Systemic Endothelial Function: Investigation of Systemic Endothelial Dysfunction in Case of Portal Hypertension Associated With Cystic Fibrosis.
Brief Title: Portal Hypertension and Systemic Endothelial Function
Acronym: ENDOTH-MUCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/33; 2015-A01872-47 (Other: ANSM)
Record Dates: First submitted 2016-06-16; First posted 2016-08-01 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Cystic Fibrosis; Portal Hypertension
MeSH Terms: conditions — Cystic Fibrosis; Hypertension, Portal | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cystic fibrosis with portal hypertension (Experimental): Mucoviscidosis with portal hypertension. Blood sample (21ml). Hepatic elastography (Fibroscan®). Measure of endothelial function (Endopat®). Injected abdominal CT scan.
  Interventions: Other: measure of endothelial function; Biological: Blood sample; Other: Hepatic elastography; Diagnostic Test: Injected abdominal CT
- Muco without portal hypertension (Experimental): Mucoviscidosis without portal hypertension. Blood sample (21ml). Hepatic elastography (Fibroscan®). Measure of endothelial function (Endopat®). Injected abdominal CT scan.
  Interventions: Other: measure of endothelial function; Biological: Blood sample; Other: Hepatic elastography; Diagnostic Test: Injected abdominal CT
- Portal hypertension without muco (Experimental): Portal hypertension without Mucoviscidosis. Blood sample (21ml) . Hepatic elastography (Fibroscan®). Measure of endothelial function (Endopat®). Injected abdominal CT scan.
  Interventions: Other: measure of endothelial function; Biological: Blood sample; Other: Hepatic elastography; Diagnostic Test: Injected abdominal CT
- Healthy volunteers (Experimental): Healthy volunteers. Blood sample (21ml) . Hepatic elastography (Fibroscan®). Measure of endothelial function (Endopat®).
  Interventions: Other: measure of endothelial function; Biological: Blood sample; Other: Hepatic elastography

INTERVENTIONS:
Other: measure of endothelial function — Arterial tone index measured by EndoPAT®. Patient should neither eat nor drink at least 4 hours before exam and should neither smoke 3 hours before the exam.
Biological: Blood sample — 21 ml of blood to measure : hepatic workup, complete blood count (CBC), platelets, prothrombin time (PT), activated partial thromboplastin time (aPTT), C-reactive protein (CRP), lipid test, ionograms, creatinine, tissue plasminogen activator factor (tPA), plasminogen activator inhibitor-1 (PAI-1), tissue factor pathway inhibitor (TFPI), Willebrand factor, soluble thrombomodulin, blood levels of endoglin and syndecan. And level beta human chorionic gonadotropin (beta-HCG) for woman only.
Other: Hepatic elastography — Hepatic elastography by Fibrocan®. Patient should neither eat nor drink at least 2 hours before exam. 10 successive measurements are made.
Diagnostic Test: Injected abdominal CT — Patient should neither eat nor drink at least 4 hours before exam.
  The examination is not realized if an abdominal scan or an MRI was performed in the five years prior to the day of the visit.
  Arms: Cystic fibrosis with portal hypertension; Muco without portal hypertension; Portal hypertension without muco

SUMMARY:
Cystic fibrosis can affect organs other than the lungs. Liver disease affects about 30% of patients: its main manifestation is the development of portal hypertension (PHT). The pathophysiology of this comorbidity is still poorly understood. It was previously considered secondary to the formation of biliary cirrhosis but another hypothesis would be that of a primitive pathology of venous vessels may cause the gradual emergence of portal hypertension without cirrhosis. Evidence indiscutly suggest that cystic fibrosis is associated with a specific endothelial dysfunction, especially as the CFTR (Cystic Fibrosis Transmembrane conductance Regulator) protein is expressed on the surface of endothelial cells. The investigators hypothesize that liver disease related to PHT-associated cystic fibrosis is associated with systemic endothelial dysfunction.

The aim is:

To demonstrate a systemic endothelial dysfunction in patients with cystic fibrosis when associated with PHT.

To study the correlations between measures of systemic endothelial function and serum markers of endothelial dysfunction and between measures of liver stiffness and systemic endothelial function.

DETAILED DESCRIPTION:
Prospective , monocentric study, with four groups of patients:

* Patients with cystic fibrosis and PHT
* Cystic fibrosis patients without PHT
* Patients free from cystic fibrosis with PHT from other causes
* Healthy controls. One study visit, no follow-up.

During the visit the following examinations will be performed:

* Collection of a blood sample of 21 mL.
* Liver eElastography achieved through hardware FibroScan® -
* Measurement of endothelial function with Endopat®
* Contrast-enhanced tomography. Abdominal CT scan will not be performed in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years.
* Patients affiliated to a social security scheme
* Patients who have given their written consent
* Four study groups:
* Group A: Patients with cystic fibrosis (CF) with liver damage and diagnosis of CF is based on sweat test and genetic analysis). PHT diagnosis is based on tomographic criteria portal vein width superior to> 15 mm, portosystemic shunt and / or splenomegaly
* Group B: cystic fibrosis patients without PHT diagnosis is based on sweat test and genetic analysis). Absence of PHTP is predicated on tomographic of Scanner.
* Group C: Patients free of CF with PHT related to another cause. Patients followed for viral liver disease (hepatitis B or C) or idiopathic portal venous system disorder, with or without cirrhosis. The diagnosis of PHT is based on tomographic criteria portal vein width superior to> 15 mm, highlighting porto-systemic shunt, splenomegaly) and / or indirect signs namely ascitis or esophageal varices.
* Group D: Healthy controls.

Exclusion Criteria:

* Patients suffering from uncontrolled hypertension despite treatment (systolic BP> 160 mmHg);
* Patient with uncontrolled diabetes (glycated Hb measurement done during the last 3 months > 7%);
* Patients with uncorrected dyslipidemia;
* Patient suffering from a sleep apnea syndrome;
* Patients with severe coagulation disorders: PR< 50%, platelets < 30,000 / microL, current anticoagulant treatment;
* Patient with contra-indication to the injection of iodinated contrast material, including history of hypersensitivity to iodinated contrast media or renal clearance failure <50 ml / min Modification of Diet in Renal Disease (MDRD) formula
* Patients allergic to latex which contra-indicates endothelial function measurement;
* Acute pathology unresolved at the time of inclusion: respiratory exacerbation, ongoing infection, recent thrombosis;
* Smoking history> 10 pack-years;
* Vasoactive therapy that may interfere with the measurement of endothelial function and cannot be stopped 24 hours before the measurement: nitrates, beta-blockers, angiotensin converting enzyme inhibitors, calcium channel blockers, inhibitors of endothelin receptors, similar prostacyclin analog, inhibitors of phosphodiesterases;
* Pregnant and lactating women (all patients with childbearing potential will only be included if their β-human chorionic gonadotropin (β-HCG) urine test is negative;
* Patient unable to provide written consent. Patient under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial systemic function measured by EndoPAT® | 30 minutes
  To compare the systemic endothelial function between the four study groups, the arterial tone index is measured by EndoPAT®.
  The EndoPAT® is the leading medical device for noninvasive endothelial function assessment. It quantifies the endothelium-mediated changes in vascular tone, elicited by a 5-minute occlusion of the brachial artery (using a standard blood pressure cuff). When the cuff is released, the surge of blood flow causes an endothelium-dependent. Flow Mediated Dilatation (FMD). The dilatation, manifested as Reactive Hyperemia, is captured by EndoPAT® as an increase in the PAT Signal amplitude. A post-occlusion to pre-occlusion ratio is calculated by the EndoPAT® software, providing the arterial tone index.

SECONDARY OUTCOMES:
Serum levels of markers of endothelial dysfunction (tPA, thrombomodulin, Willebrandt factor, PAI1) | 30 minutes
  Blood sample (21 ml) is collected from each patients to dose the markers of endothelial dysfunction (tPA, thrombomodulin, Willebrandt factor, PAI1).
  The objective is to compare for the 4 groups the relations between:
  * the serum levels of markers of endothelial dysfunction and peripheral endothelial function;
  * And the serum levels of markers of endothelial dysfunction and the presence of portal hypertension (HTP).
Endogline/Syndecan-4 ratio measurement | 30 minutes
  Blood sample (21 ml) is collected from each patients to measure the blood levels of endoglin and syndecan.
  Endoglin and syndecan-4 are transmembrane glycoproteins present on endothelial cells.
  The objective is to compare for the 4 group the relation between :
  * endoglin/syndecan-4 ratio and peripheral endothelial function;
  * and, endoglin/syndecan-4 ratio and presence of HTP.
Measurement of hepatic elasticity by Fibroscan® | 30 minutes
  The objective is to compare for the 4 groups the relations between hepatic elasticity and endothelial systemic function.
  The Fibroscan measures the velocity of the sound wave passing through the liver from the device and then converts that measurement into a liver elasticity measurement. The result reveals the health of the liver: more the liver is hard, more his state is pathologic.
Hepatic abnormalities observed on injected abdominal CT. | 30 minutes
  All hepatic abnormalities observed on injected abdominal CT for groups A, B and C are analyzed.
  The objective is to compare the hepatic radiologic abnormalities associated with HTP in cystic fibrosis with hepatic radiologic abnormalities associated with HTP from other causes.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Grenet, MD, Principal Investigator — Hopitral Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No